CLINICAL TRIAL: NCT06859671
Title: A Randomized Study of a Short Duration Therapy for Candidemia
Acronym: CANDISHORT
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP230824
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: CANDIDEMIA
MeSH Terms: conditions — Candidemia | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Design of the study Multicenter, controlled, randomized, non-inferiority, clinical trial with 2 parallel groups (1:1)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 14 days of antifungal treatment (Active Comparator)
  Interventions: Drug: Standard of Care (SOC)
- 7 days of antifungal treatment (Experimental)
  Interventions: Drug: Shortened duration of antifungal therapy

INTERVENTIONS:
Drug: Standard of Care (SOC) — 14 days of antifungal therapy after the 1st negative blood culture
  Arms: 14 days of antifungal treatment
Drug: Shortened duration of antifungal therapy — 7 days of antifungal therapy after the 1st negative blood culture
  Arms: 7 days of antifungal treatment

SUMMARY:
Scientific justification Candidemia is a major public health problem. In France, the 30-day mortality of candidemia varies from 30% to 50% depending on the need for intensive care and it has not decreased in 30 years.

The duration of treatment for candidemia was set at a minimum of 14 days after the last positive blood culture following the Rex trial (1) comparing the efficacy of fluconazole vs amphotericin B where the minimum duration of treatment was imposed. The risk of a too short treatment is the absence of control of the candidemia with secondary dissemination, in particular cardiac and ophthalmic.

A retrospective study looking at the risk of ophthalmologic complications after candidemia found among the 21/78 treated for less than 14 days, only one case of late endophthalmitis in a patient who had only been treated for 48 hours. In addition, the prolonged duration of antifungals exposes the risk of selection of more resistant strains with a modification of the flora, with the possibility of acquiring resistance as early as 8 days of treatment with caspofungin, and has a greater liver toxicity.

There is no prospective study on the direct impact of antifungal agents (type of antifungal agent and duration) on the mycobiota.

ELIGIBILITY:
Inclusion Criteria:

* Adults (Age ≥ 18 years old)
* With an uncomplicated candidemia defined by the absence of secondary sites requiring prolonged treatment: endocarditis, ophthalmologic involvement, thrombosed catheter, arthritis, meningitis, candida abscess that cannot be drained, pyelonephritis.
* Without expected aplasia duration greater than 7 days
* Being apyretic and having a 1st negative blood culture after diagnosis
* Removal of the vascular catheter if present
* Written informed consent from the patients or his/her relatives
* Patients with less than 7 days of aplasia predictable

Exclusion Criteria:

* Presence of an indwelling vascular catheter or device that cannot be removed or an abscess that cannot be drained and is likely to be the source of candidemia or the presence of secondary sites of candidemia requiring prolonged treatment
* Patients with more than 7 days of aplasia
* Candida strain resistant to the antifungal used
* Pregnancy, breastfeeding
* Hypersensitivity or previous severe adverse drug reaction to the antifungal treatments.
* unwilling, in the judgment of the investigator, to comply with the protocol
* Patient under legal guardianship or without healthcare coverage
* Women with childbearing potential not using adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality (ACM) | At day 28
  at day 28 after the 1st negative blood culture under antifungal treatment for all patients included with an uncomplicated candidemia

SECONDARY OUTCOMES:
Proportion of patients with secondary localizations | At day 28
Cumulative incidence of death related to fungal infection | At day 28
  at Day 28 after the 1st negative blood culture under antifungal treatment
Aspartate Amino-transferase level | At day 14
Aspartate Amino-transferase level | At day 28
alanine aminotransférase (ALAT) level | At day 14
alanine aminotransférase (ALAT) level | At day 28
Gamma-Glutamyl Transférase (GGT) level | At day 14
Gamma-Glutamyl Transférase (GGT) level | At day 28
Bilirubin blood levels | At day 14
Bilirubin blood levels | At day 28
Cost per extra-day alive without antifungal treatment | Up to day 28
  Incremental cost effectiveness ratio

IPD SHARING:
Plan to Share IPD: Undecided